CLINICAL TRIAL: NCT07069985
Title: Assessment of Sexual Function in Male Patients Undergoing Hydrocelectomy and Their Partners: A Prospective Study Based on IIEF an FSFI Scores
Brief Title: Assessment of Sexual Function in Male Patients Undergoing Hydrocelectomy and Their Partners
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: University of Health Sci ATRH; Secondary ID: 756 (Other: UHS, Ankara Training and Research Hospital Ethics Committee)
Record Dates: First submitted 2025-06-11; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-05

CONDITIONS: Hydrocelectomy; Erectile Dysfunction; Sexual Dysfunction Male; Sexual Dysfunction Female
Keywords: erectile dysfunction; hydrocelectomy; sexual dysfunction
MeSH Terms: conditions — Erectile Dysfunction; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: male patients who underwent hydrocelectomy, group 2: partners of the male patients: Group 1: Heterosexual male patients who underwent hydrocelectomy in our clinic between 2020 and 2024. Sexually active patients between the ages of 18-75 years who underwent hydrocelectomy and who had no previous history of scrotal surgery were included. Patients with postoperative complications (large scrotal hematoma), those with mental or physical disabilities, and those with preoperative moderate to severe erectile dysfunction were excluded.
  Group 2: Female partners of the male patients who underwent hydrocelectomy.

SUMMARY:
This study aimed to assess changes in sexual function in men undergoing hydrocelectomy and their partners.

Male patients who underwent hydrocelectomy in our clinic between 2020 and 2024 were included in the study This study was designed as a prospective cohort. Sexually active male patients between the ages of 18 and 75 who underwent hydrocelectomy and had no history of previous scrotal surgery were included. Patients with postoperative complications such as large scrotal hematomas, mental or physical disabilities, or moderate to severe erectile dysfunction before surgery were excluded. Written informed consent was obtained from both the patients and their partners.

Demographic and clinical data including age, comorbidities, previous surgeries, and the presence of penile abnormalities were recorded. Penile length was measured in a temperature-controlled room (23-25°C) under similar conditions for all patients. Measurements were taken in the flaccid state, from the base to the tip along the dorsal side, using a ruler marked in millimeters by the same physician. The size of the hydrocele was also recorded: the largest vertical diameter (top to bottom) was defined as the vertical size, and the largest horizontal diameter (side to side) as the transverse size.

Sexual function was assessed through face-to-face interviews, with attention to social distancing. Questionnaires were administered before surgery and again one month after the operation. Male patients completed the International Index of Erectile Function (IIEF), which includes 15 items and a total possible score of 75, covering five domains: erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction. Female partners were evaluated using the Female Sexual Function Index (FSFI), consisting of 19 items and six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain, with a maximum score of 36.

A post hoc power analysis was performed using G*Power 3.1.9.7. Based on an effect size of 0.5 and a significance level of 0.05, a sample size of 44 was calculated to provide 90% power. Statistical analysis was conducted using IBM SPSS version 20. Normality was checked using the Shapiro-Wilk test and P-P plots. Normally distributed data were presented as mean ± standard deviation, while non-normally distributed data were expressed as median (minimum-maximum). Categorical variables were shown as numbers and percentages. The Pearson Chi-square test was used for comparing categorical variables. The paired samples t-test was used to compare pre- and postoperative scores of the sexual function questionnaires. A p-value of less than 0.05 was considered statistically significant.

DETAILED DESCRIPTION:
We hypothesized that men who underwent hydrocelectomy and their partners would have improved sexual function in the postoperative period compared to the preoperative period. In our study, we aimed to compare preoperative and postoperative sexual dysfunction in 80 male patients who underwent hydrocelectomy and their partners using nationally validated sexual function assessment questionnaires.

Male patients who underwent hydrocelectomy in our clinic between 2020 and 2024 were included in the study. The study was designed as a prospective cohort. Sexually active patients between the ages of 18-75 years who underwent hydrocelectomy and who had no previous history of scrotal surgery were included. Patients with postoperative complications (large scrotal hematoma), those with mental or physical disabilities, and those with preoperative moderate to severe erectile dysfunction were excluded. Written informed consent was obtained from all patients and their partners. Patients' age, comorbidities, previous operations and presence of penile anomalies were reported. Penile length was measured under similar environmental conditions (air-conditioned room and temperatures ranging from 23 to 25°C). The penis was measured from the base to the distal tip in the flaccid state by the same physician along the penile dorsum with a millimeter-marked ruler. The largest diameter between the top and bottom of the hydrocele sac was measured and reported as vertical hydrocele size, and the largest diameter between lateral and medial was measured and reported as transverse hydrocele size by the same physician.

Assessment of sexual function All patients and their partners were interviewed face-to-face, social distancing rules were observed and sexual function assessment questionnaires were administered. The questionnaires were administered preoperatively and at 1 month postoperatively. For male patients, the nationally validated International Index of Erectile Function (IIEF) questionnaire consisting of 15 questions with a maximum total score of 75 was administered. This questionnaire includes 5 subgroups: erectile function, orgasmic function, sexual desire, sexual satisfaction and overall satisfaction (8). Female partners were assessed using the Female Sexual Function Index (FSFI), which consists of 19 questions and has a maximum total score of 36. This questionnaire includes 6 subgroups: sexual desire, sexual arousal, lubrication, orgasm, satisfaction and pain (9).

Statistical Analysis Post Hoc Power analysis was performed. (G*Power 3.1.9.7 software, Heinrich-Heine-Universität Düsseldorf, Düsseldorf, Germany). When the effect size was taken as 0.5 and the study power was calculated as 90%, the number of patients required for the study was calculated as 44 with a margin of error of 0.05.

While evaluating the data obtained in the study, IBM SPSS (Statistical Package for the Social Sciences) program version 20 was used for statistical analysis (SPSS, Chicago, IL). Shapiro-Wilk and P-P plot analysis were used to test the conformity of continuous data to normal distribution. Data conforming to normal distribution were reported as mean ± standard deviation (SD) and data not conforming to normal distribution were reported as median (minimum-maximum). Categorical data were given as number and percentage (%) and Pearson Chi-square test was used to compare categorical data between groups. Paired samples t-test was used to compare preoperative and postoperative sexual function assessment questionnaires and subgroups. All statistical tests were two-tailed and p<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active patients between the ages of 18-75 years who underwent hydrocelectomy and who had no previous history of scrotal surgery were included.

Exclusion Criteria:

* Patients with postoperative complications (large scrotal hematoma), those with mental or physical disabilities, and those with preoperative moderate to severe erectile dysfunction were excluded.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male patients who underwent hydrocelectomy in our clinic between 2020-2024 and their partners
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Changes in International Index of Erectile Function (IIEF) questionnaire | 1 month after hydrocelectomy
  The questionnaires were administered preoperatively and at 1 month postoperatively. For male patients, the nationally validated International Index of Erectile Function (IIEF) questionnaire consisting of 15 questions with a maximum total score of 75 was administered. This questionnaire includes 5 subgroups: erectile function, orgasmic function, sexual desire, sexual satisfaction and overall satisfaction.
Changes in Female Sexual Function Index (FSFI) | 1 month after hydrocelectomy
  The questionnaires were administered preoperatively and at 1 month postoperatively. Female partners were assessed using the Female Sexual Function Index (FSFI), which consists of 19 questions and has a maximum total score of 36. This questionnaire includes 6 subgroups: sexual desire, sexual arousal, lubrication, orgasm, satisfaction and pain. Increases in total IIEF and its subdomain scores, as well as in total FSFI and the subdomains of desire, arousal, lubrication, orgasm, and satisfaction, indicate improvement; an increase in the FSFI pain score reflects reduced pain.

CONTACTS AND LOCATIONS:
Overall Officials: Omer G Doluoglu, Professor, Study Director — UHS, Department of Urology Clinic of Ankara Training and Research Hospital
Locations (1):
- University of Medical Sciences, Department of Urology Clinic of Ankara Training and Research Hospital, Ankara, Turkey (Türkiye)